CLINICAL TRIAL: NCT02302443
Title: A First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single Administration of HM12470 in Subjects With Type 1 (T1DM) and Type 2 Diabetes Mellitus (T2DM)
Brief Title: A First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM12470
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-INS115-101
Record Dates: First submitted 2014-11-19; First posted 2014-11-27 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): Very low dose of HM12470 (single dose, subcutaneous injection)
  Interventions: Biological: HM12470
- Cohort 2 (Experimental): Low dose of HM12470 (single dose, subcutaneous injection)
  Interventions: Biological: HM12470
- Cohort 3 (Experimental): Intermediate dose of HM12470 (single dose, subcutaneous injection)
  Interventions: Biological: HM12470
- Cohort 4 (Experimental): High dose of HM12470 (single dose, subcutaneous injection)
  Interventions: Biological: HM12470
- Cohort 5 (Experimental): Active comparator and a selected dose of HM12470 (single dose, subcutaneous injection)
  Interventions: Biological: HM12470; Biological: Active comparator
- Cohort 6 (Experimental): Active comparator and a selected dose of HM12470 (single dose, subcutaneous injection)
  Interventions: Biological: HM12470; Biological: Active comparator

INTERVENTIONS:
Biological: HM12470 — Single dose subcutaneous administration ranging from a very low dose to high dose
Biological: Active comparator — Single dose subcutaneous administration of active comparator
  Arms: Cohort 5; Cohort 6

SUMMARY:
The purpose of this study is to investigate safety, tolerability, pharmacokinetics (PK) ad pharmacodynamics (PD) of HM12470 after single injection in T1DM and T2DM patients.

DETAILED DESCRIPTION:
This study is designed to evaluate safety, tolerability, PK and PD of HM12470 after single administration in subjects with T1DM and T2DM. In some cohorts for this study, the safety, tolerability, PK and PD of HM12470 will be compared with that of commercially available insulin.

ELIGIBILITY:
Inclusion Criteria for T1DM:

* T2DM more than 12 monthM
* Age ≥18 and ≤70 years
* Body mass index between 18.0 and 35.0 kg/m2 inclusive.
* Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
* Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or post-menopausal for >12 months. Males must be surgically sterile, abstinent or if engaged in sexual relations of child-bearing potential, the subject must be using an acceptable contraceptive method during and for during a period of 60 days after the last dose of Study Drug.
* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject).

Inclusion Criteria for T2DM:

* T1DM more than 12 monthM
* Age ≥18 and ≤70 years
* Body mass index between 18.0 and 30.0 kg/m2 inclusive.
* Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
* Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or post-menopausal for >12 months. Males must be surgically sterile, abstinent or if engaged in sexual relations of child-bearing potential, the subject must be using an acceptable contraceptive method during and for during a period of 60 days after the last dose of Study Drug.
* Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject).

Exclusion Criteria

* A subject who has proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator
* Recurrent major hypoglycemia or hypoglycemic unawareness or recent ketoacidosis
* pregnant or lactating women
* participation in an investigational study within 30 days prior to dosing
* Clinically significant abnormal ECG at screening, as judged by the Investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events | 1 month

SECONDARY OUTCOMES:
Peak Plasma Concentration(Cmax) of HM12470 following a single dose | 1 month
  Pharmacokinetic properties of HM12470 following a single dose will be assessed in plasma using a validated assay
Area under the concentration-time curve (AUC) of HM12470 following a single dose | 1 month
  Pharmacokinetic properties of HM12470 following a single dose will be assessed in plasma using a validated assay

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Pharmaceuticals Hanmi Pharmaceuticals, Study Director — Hanmi Pharmaceuticals
Locations (1):
- Hanmi Pharmaceutical Company, Seoul, South Korea